CLINICAL TRIAL: NCT04202003
Title: A Multicenter, Open-label, Phase 1/2a Study to Evaluate the Safety and Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of TJ011133 as Monotherapy and in Combination With Azacitidine (AZA) in Patients With Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)
Brief Title: A Study to Evaluate the Safety and Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of TJ011133 as Monotherapy and in Combination With Azacitidine (AZA) in Patients With Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TJ Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ011133AML102
Record Dates: First submitted 2019-12-13; First posted 2019-12-17 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndromes(MDS)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TJ011133 (Experimental): This is an open-label Phase 1/2a clinical study. The study will be conducted in two parts: Part I: Phase 1 dose escalation, TJ011133 is tentatively scheduled to be administered once weekly in 28-day treatment cycles;Part II: Phase 2a study TJ011133 will be administered at a dose of 30 mg/kg once weekly, and AZA will be administered at a dose of 75 mg/m2 by subcutaneous injection for 7 consecutive days from D1 to D7 in 28-day treatment cycles.
  Interventions: Drug: TJ011133

INTERVENTIONS:
Drug: TJ011133 — This is an open-label Phase 1/2a clinical study. The study will be conducted in two parts: Part I: Phase 1 dose escalation, TJ011133 is tentatively scheduled to be administered once weekly in 28-day treatment cycles;Part II: Phase 2a study TJ011133 will be administered at a dose of 30 mg/kg once weekly, and AZA will be administered at a dose of 75 mg/m2 by subcutaneous injection for 7 consecutive days from D1 to D7 in 28-day treatment cycles.

SUMMARY:
This study is a phase I/II study of TJ011133 as Monotherapy and in Combination with Azacitidine (AZA) in Patients with Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS). This study include Phase I and Phase IIa study. Phase I study ClinicalTrials.gov ID is NCT04202003 and this is for phase IIa study. Phase IIa study is designed to preliminarily assess the efficacy and safety of TJ011133 in combination with AZA as first-line treatment in patients with newly diagnosed AML who are intolerant to standard induction chemotherapy or patients with treatment naive, intermediate and high-risk MDS.

ELIGIBILITY:
Inclusion Criteria

Phase 1 single dose escalation:

* Male or female, aged ≥ 18 and ≤ 70 years at the time of signing informed consent form;
* For the disease under study, enrollment may be considered if one of the following is satisfied:

  1. Subjects must be with pathologically diagnosed as acute myeloid leukemia (AML) according World Health Organization (WHO) 2016 classification criteria, with the exception of acute promyelocytic leukemia; it is a recurrent or refractory disease without other available appropriate conventional treatments;
  2. Subjects with intermediate- and high-risk relapsed/refractory MDS (IPSS-R score >3.5) who are pathologically confirmed and meeting the diagnostic criteria of World Health Organization (WHO) 2016 or who are unable to tolerate the treatment of demethylation drugs or other drugs (e.g., treatment-emergent Grade 3 or higher drug-related hepatic and/or renal toxicities leading to permanent withdrawal during treatment), and the investigator judges that there is no other appropriate treatment;
* For patients with MDS, a blast percentage of < 20% is required in bone marrow aspiration smear or bone marrow biopsy pathology at screening;
* ECOG score 0-2;
* Subjects have been recovered from the toxicity of previous anti-AML/MDS treatments (according to NCI CTC AE 5.0 ≤ Grade 1, except alopecia) ;
* Subjects must have adequate liver function, renal function and coagulation function. The laboratory tests within 7 days before the first dose should meet the following requirements:

  1. Liver function:

     * Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN);
     * AST and ALT ≤ 2.5 × ULN.
  2. Renal function:

     -Serum creatinine ≤ 1.5 × ULN or estimated creatinine clearance ≥ 50 mL/min according to the Cockcroft-Gault equation (Appendix 5).
  3. Coagulation function:

     * International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN;
     * Activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN.

Subjects for Phase 2a combination therapy:

* Male or female, aged ≥ 18 years at the time of signing informed consent form;
* For the disease under study, enrollment may be considered only if the following conditions are met:

Newly diagnosed AML with intolerance to standard induction chemotherapy/intermediate- and high-risk (International Prognostic Scoring System IPSS-R) MDS (only applicable for Phase 2a study); symptomatic treatment such as hydroxycarbamide, erythropoietin, and/or hematopoietic growth factors are allowed within 7 days of the first dose;

* The subject's ECOG score has to meet the following criteria:

  * Newly diagnosed AML with intolerance to standard induction

    * Newly diagnosed intermediate- and high-risk MDS: ECOG score 0 - 2
* Subjects must have adequate liver function, renal function and coagulation function. The laboratory tests within 7 days before the first dose should meet the following requirements::

  1. Liver function:

     * Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN); total bilirubin ≤ 3 × ULN is allowed for subjects aged 18 - 74 years (only for newly diagnosed AML subjects who are intolerant to standard induction chemotherapy)
     * AST and ALT ≤ 3 × ULN.
  2. Renal function:

     -Estimated creatinine clearance ≥ 50 mL/min according to the Cockcroft-Gault equation (Appendix 5); creatinine clearance ≥ 30 mL/min is allowed for subjects aged 18 - 74 years (only for newly diagnosed AML subjects who are intolerant to standard induction chemotherapy)
  3. Coagulation function:

     * International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN;
     * Activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN.

All subjects:

* Expected survival ≥ 12 weeks;
* White blood cell count (WBC) ≤ 25 × 103/μL within 7 days prior to the first dose (hydroxycarbamide or leukapheresis is allowed to meet this criterion);
* Subjects must be willing to provide available diagnostic evidence or undergo bone marrow aspiration and biopsy before study treatment, and must be willing to undergo bone marrow aspiration and biopsy after receiving study treatment;
* Subjects must give informed consent before starting the study and sign written consent voluntarily by themselves (or their legal representatives). Subjects or their legal representatives should be able to communicate well with investigators and agree to adhere with the study protocol and complete the study.

Exclusion Criteria

Phase 1 single dose escalation:

* Previously received treatment with other drug therapies targeting CD47;
* Previously received CAR-T cell therapy;
* Previously received treatment with PD1 or PDL1 antibody;
* Previously received or planned to receive allogeneic stem cell transplantation during the study, or autologous stem cell transplantation within 3 months prior to the first dose of study drug;
* Subjects have received chemotherapy, immunotherapy, radiotherapy, major surgery within 4 weeks prior to the first dose;
* Subjects' cardiac function meet any of the following criteria:

  * Subjects have any kind of clinically significant rhythm abnormalities or conduction abnormalities that require clinical intervention;
  * Subjects have congenital QT prolongation syndrome or QTc > 450 msec in men, QTc > 470 msec in women (QTc calculated using Fridericia's correction formula [Appendix 6]), or on medications that may cause QT prolongation or torsades de pointes;
  * Subjects have any kind of clinically significant cardiovascular diseases, including acute myocardial infarction, unstable angina, coronary artery bypass surgery or peripheral artery bypass surgery, cerebrovascular events (thromboembolic or hemorrhagic cerebrovascular events, excluding transient ischemic attack), New York Heart Association (NYHA) (Appendix 7) ≥ Grade 3 congestive cardiac failure, or left ventricular ejection fraction (LVEF) < 40% within 3 months prior to enrollment; Phase 2a combination therapy
* Previously received treatment with demethylated drugs or cytotoxic drugs in patients with MDS;
* Previously received any anti-tumor therapy for AML;
* AML with a good prognosis, including cytogenetic alterations, such as t (8;21), inv (16) or t (16;16) or t (15;17);
* Subjects are known to have allergy to AZA or mannitol;
* Subjects' cardiac function meet any of the following criteria:

  * Subjects have any kind of clinically significant rhythm abnormalities or conduction abnormalities that require clinical intervention;
  * Subjects have congenital QT prolongation syndrome or taking drugs that may cause QT prolongation or torsades de pointes;
  * Subjects have any kind of clinically significant cardiovascular diseases, including acute myocardial infarction, unstable angina, coronary artery bypass surgery or peripheral artery bypass surgery, cerebrovascular events (thromboembolic or hemorrhagic cerebrovascular events, excluding transient ischemic attack), New York Heart Association (NYHA) (Appendix 7) ≥ Grade 3 congestive cardiac failure within 3 months prior to enrollment;
* Subjects have undergone major surgery within 4 weeks prior to the first dose;

All subjects:

* Subjects have received vaccination within 4 weeks prior to the first dose and/or planned vaccination after participating in the study;
* Subjects have received clinical trial drug treatment within 4 weeks prior to the first dose or currently participating in other interventional clinical trials;
* Subjects are known to have hereditary or acquired hemorrhagic disorders;
* Subjects have hypertension uncontrollable with drug therapy (systolic blood pressure ≥ 140 mmHg, or diastolic blood pressure ≥ 90 mmHg at rest);
* Subjects suffer from disease that requires long-term use of systemic steroid therapy or other immunosuppressive therapy. However, subjects who use physiologic replacement doses of hydrocortisone or drugs of equivalent doses (Appendix 8), i.e., up to 20 mg of hydrocortisone (or 5 mg of prednisone) in the morning and up to 10 mg of hydrocortisone (or 2.5 mg of prednisone) at night, may be considered for enrollment;
* Subjects are known to have central nervous system (CNS) involvement;
* Subjects are known to have HIV infection (anti-HIV positive), active hepatitis B (HBsAg positive, or HBcAb positive and HBV-DNA PCR positive), or active hepatitis C (anti-HCV antibody positive and HCV-RNA PCR positive), or syphilis infection (anti-TP test positive);
* Subjects have a history of solid organ transplantation;
* Subjects plan to receive other anti-tumor therapies, including but not limited to chemotherapy, biotherapy, immunotherapy, hormone therapy and traditional Chinese medicine, while participating in the study;
* Subjects have a history of autoimmune disease or active autoimmune disease;
* Subjects have uncontrolled active infection;
* Subjects have severe electrolyte disturbances that cannot be corrected;
* Subjects have a history of other malignancies, except for clinically cured malignancies (no relapse for at least 5 years), cured carcinoma in situ, and skin cancer other than malignant melanoma;
* Subjects have a history of psychotropic drug abuse and are unable to quit or have mental disorders, or have concomitant diseases that seriously endanger patients' safety or hinder the study completion at the discretion of investigators;
* Subjects are women during pregnancy or lactation, or women and men with fertility planning;
* The investigators consider that patients have other factors that may affect the results of the study and interfere with their full participation in the study, including previous or existing health conditions or medical or laboratory abnormalities, or put them at high risk.
* Subjects with MDS who meet any of the following must also be excluded:
* Subjects have uncorrected serum folic acid deficiency or vitamin B12 deficiency;
* MDS transformed from previously existing myeloproliferative tumors (MPN) or MDS/MPN types conforming to WHO 2016 classification standard include chronic myelomonocytic leukemia (CMML), atypical chronic myeloid leukemia (aCML), juvenile myelomonocytic leukemia (JMML), etc..

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities(DLT) | 28days after first dose
  To evaluate the safety and tolerance of TJ011133 monotherapy in patients with r/r AML or MDS
Maximum tolerable dose(MTD) | Through study completion, an average of 1 year
  To explore the maximum tolerable dose (MTD) of TJ011133 monotherapy for patients with r/r AML or MDS, the recommended phase II dose (RP2D) and the optimal dosage regimen.
Recommended phase II dose | Through study completion, an average of 1 year
  Recommended phase II dose (RP2D)
Complete response rate (CR rate) only for phase 2a | Through study completion，an average of 1 year
  Preliminary efficacy endpoints (only for Phase 2a): for response assessment in AML/MDS patients, the complete response rate (CR rate) will be evaluated according to the ELN2017/IWG 2006 criteria

CONTACTS AND LOCATIONS:
Locations (26):
- China (26):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality
  - Beijing Boren Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Zhujiang Hospital Of Southern Medical University, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Second Hospital of HeBei Medical University, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Suzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Xi'an Jiaotong University（Xibei Hospital）, Xi’an, Shanxi
  - Institute of Hematology and Blood Disease Hospital, Chinese Academy of Medical, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No